CLINICAL TRIAL: NCT06263374
Title: Effect of Maxillofacial Physiotherapy With Addition of Motor Imagery vs Sham on the Recovery of Mobility, Jaw Function, and Quality of Life After Orthognathic Surgery: A Single-Blind Randomized Controlled Study
Brief Title: Maxillofacial Rehabilitation Using Motor Imagery vs Sham After Orthognathic Surgery
Acronym: MAXIMAND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 69HCL21_0355
Record Dates: First submitted 2024-02-01; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Maxillofacial Abnormalities
Keywords: Motor imagery; Maxillofacial physiotherapy; Orthognathic surgery
MeSH Terms: conditions — Maxillofacial Abnormalities

STUDY DESIGN:
Intervention Model Description: Multi-centric randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: A randomization list will be centrally generated by an independent methodologist for each center and integrated into the electronic case report form. The physiotherapist will disclose the allocation to the participant during the inclusion visit, following clear, transparent, and appropriate information, and obtaining the participant's consent to participate in the study. This disclosure occurs after all measurements have been completed. The inclusion visit is scheduled 30 days ± 8 before the surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy with self-rehabilitation including motor imagery (Experimental): Patients will undergo maxillofacial rehabilitation, comprising a single 30-minute session per week during the first month post-surgery, followed by one session every two weeks for up to three months. In between these sessions, patients will participate in a self-rehabilitation program at home, involving jaw and tongue movements as well as massages, each lasting 5 minutes, three times a day. Compliance with the program will be monitored by the physiotherapist. The program has been standardized across all centers, ensuring consistency in this multicentric study.
  Interventions: Behavioral: Motor imagery of the jaw
- Physiotherapy with self-rehabilitation including control task (Sham Comparator): Patients allocated to the control group will receive physiotherapy along with self-rehabilitation, incorporating a control task. The delivery of physiotherapy and self-rehabilitation will mirror that of the experimental group. The control task, substituting motor imagery, will involve completing Sudoku or crossword puzzles based on patient preference. (i.e., an equivalent duration to the motor imagery practice of the experimental group). The physiotherapist will ensure adherence to the rehabilitation and intervention protocols.
  Interventions: Behavioral: Control task (Sudoku or Crossword puzzle)

INTERVENTIONS:
Behavioral: Motor imagery of the jaw — Fifty individuals who have undergone orthognathic surgery of the mandible alone or concurrently with the maxilla will be randomly assigned to the experimental group, which involves practicing motor imagery in addition to a self-rehabilitation program and physiotherapy. Patients will be guided to visualize three sets of jaw movements three times a day. Adherence to the program will be monitored by the physiotherapist. The program has been standardized across all participating centers as the study is multicentric.
  Arms: Physiotherapy with self-rehabilitation including motor imagery
Behavioral: Control task (Sudoku or Crossword puzzle) — Fifty individuals who have undergone orthognathic surgery of the mandible alone or concurrently with the maxilla will be randomly assigned to the control group, which involves practicing a control task (completion of Sudoku or crossword puzzles) in addition to a self-rehabilitation program and physiotherapy. Patients will be instructed to engage in the task for approximately 10 minutes per day, equivalent to the duration of motor imagery practice in the group 1. Adherence to the program will be monitored by the physiotherapist. The program has been standardized across all participating centers, as the study is multicentric.
  Arms: Physiotherapy with self-rehabilitation including control task

SUMMARY:
Dento-maxillary dysmorphoses are defined as an anomaly in the relative growth of the maxilla and/or mandible. They lead to functional disorders (i.e., disturbances in chewing or oral communication) and aesthetic issues with psychological repercussions on self-esteem, affecting the quality of life of these patients. The multidisciplinary treatment involves orthodontics (duration = 18-24 months), orthognathic surgery involving the maxillary and/or mandibular bone (at 12 months), immediately followed by physiotherapy (duration = 3 months). One main goal after surgery is the recovery of month opening to restore an appropriate orofacial function. Motor imagery (mental rehearsal of a movement without actually moving) is effectively used in athletes and in rehabilitation mainly neurological but so far has not been investigated in maxillofacial rehabilitation. Considering that the effectiveness of rehabilitation is increased when physical and mental practices are combined, this leads to propose this study aiming to investigate whether the addition of motor imagery of the maxillofacial region to maxillofacial physiotherapy (based on a practice of physical therapeutic exercises) modifies the recovery of maximum mouth opening, other ranges of motion, jaw function, and quality of life in patients after orthognathic surgery compared to the addition of a control cognitive task [watching a non-emotional content film or filling out a crossword or Sudoku grid] to maxillofacial physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer after orthognathic surgery of the mandible alone or concurrently with the maxilla.
* Consent to participate to the study after receiving clear, loyal and appropriate information.
* Aged ≥ 18 years.
* Health care beneficiary

Exclusion Criteria:

* Patient who has undergone maxillary surgery alone (e.g., LeFort I) or genioplasty. Indeed, both of these surgeries typically have a favorable and rapid recovery without the need for maxillofacial physiotherapy.
* Patient unable to imagine a maximum mouth opening movement (i.e., score = 1, no mental image / no sensations) on the 5-point Likert scale used during the administration of the Tongue Month Imagery Questionnaire (TMIQ).
* Ongoing participation in another research that aim to evaluate an intervention likely to improve the neurological or functional recovery introducing an experimental bias.
* Patients not undergoing rehabilitation in the study centers.
* Patients under guardians, curators, or legal protection.
* Pregnant or lactating patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Maximal mouth opening measured in millimeters using a caliper | Day 30
  Active range of motion for maximum mouth opening in millimeters measured using a caliper between the maxillary and mandibular incisors on the midline. This measure has an excellent reliability (Best et al., 2013), including in case of orthognathic surgery (Ellis et al., 1989) (Ueki et al., 2008). The minimum clinical change is 5 mm for patients experiencing a reduction in maximum mouth opening due to pain (Kropmans et al., 1999). This measurement will be performed by an evaluator blinded to the randomization group.

SECONDARY OUTCOMES:
Active maximum mouth opening in millimeter using a vernier caliper | Day 0 ; Day 7 ; Day 14 ; Day 21 ; Day 30 ; Day 45 ; Day 60 ; Day 75 ; Day 90 ; Day 180
  Compare active maximum mouth opening in millimeter obtained using a vernier caliper between the experimental group (i.e., motor imagery of the maxillofacial region [MI maxillofacial] + maxillofacial physiotherapy) and the control group (control cognitive task [watching a non-emotional content film or filling out a crossword or Sudoku grid] + maxillofacial physiotherapy), taking into account the possibility of orthodontic treatment with prescribed and effectively worn retention elastics.
Active jaw range of motion (ROM) other than maximal opening | Day 0 ; Day 7 ; Day 14 ; Day 21 ; Day 30 ; Day 45 ; Day 60 ; Day 75 ; Day 90 ; Day 180
  Active range of motion for maximum mouth opening in millimeters measured using a caliper between the maxillary and mandibular incisors on the midline. Forward and lateral jaw movements will be measure by the same evaluator blinded to the randomization group.
Maxillofacial pain | Day 0 ; Day 7 ; Day 14 ; Day 21 ; Day 30 ; Day 45 ; Day 60 ; Day 75 ; Day 90 ; Day 180
  Pain at rest and during jaw movements will be assessed using the 0-100mm Visual Analog Scale (VAS) (0=no pain, 100=maximum imaginable pain). In the evaluation of acute pain, the Visual Analog Scale is commonly used as it is a reliable, valid, sensitive, and suitable measurement tool (Sirintawat et al., 2017). Analgesic consumption will be recorded through patient inquiry at each physiotherapy session.
Body weight mass (kilograms) | Day 0 ; Day 7 ; Day 14 ; Day 21 ; Day 30 ; Day 45 ; Day 60 ; Day 75 ; Day 90 ; Day 180
  The patient will be weighed using a scale at the end of each physiotherapy session.
Orthodontic associated treatment | Day 0 ; Day 7 ; Day 14 ; Day 21 ; Day 30 ; Day 45 ; Day 60 ; Day 75 ; Day 90 ; Day 180
  Orthodontic treatment concurrent with physiotherapy will be systematically assessed at each physiotherapy session by questioning the patient, including an inquiry about any prescribed orthodontic measures and the use of retention elastics, as these factors may impact the maximum mouth opening.
Compliance with physiotherapy and intervention | Day 7 ; Day 14 ; Day 21 ; Day 30 ; Day 45 ; Day 60 ; Day 75 ; Day 90
  This will include i) the physiotherapy number (n=8) and duration (each session duration = 30 min), ii) the compliance with active movement performed self-rehabilitation (both motor imagery control groups) indicated by the number of movement practiced per day, iii) compliance with intervention (motor imagery or control). The physiotherapist will supervised and verify the patient's compliance all along the study.
Orofacial function | Day-30 ; Day 30 ; Day 90 ; Day 180
  It will be measured using the Jaw Functional Limitation Scale 8 items. The patient will rate each item from 0 (no discomfort) to 10 (complete limitation). The maximum total score is 80. This scale includes items specifically assessing chewing, vertical jaw mobility, as well as verbal and emotional expression. The questionnaire is reliable (Ohrbach, Larsson, et al., 2008).
Maxillofacial quality of life | Day-30 ; Day 30 ; Day 90 ; Day 180
  It will be measure using the Orthognathic Quality of Life Questionnaire with 22 items. Each item is assessed from 0=no discomfort to 4=major discomfort, with a maximum total score of 88. Four sub-domains are evaluated: aesthetics (max subscore=20, items 1, 7, 10-11, 14), function (max subscore=20, items 2-6), awareness of facial deformity (max subscore=16, items 8-9, 12-13), and social impact (max subscore=32; items 15 to 22) (Cunningham et al., 2000).
Level of achievement of the goals set by the patient before surgery | Day-30 ; Day 90 ; Day 180
  We will use the Goal Attainment Scale (Krasny-Pacini et al., 2013). Before surgery, the patient will choose the 3 items that they consider to be the most critical/disturbing among the various domains impacted by dento-maxillary dysmorphosis, The patient will indicate the level of achievement for each of these goals [initial pre-treatment level = -2 ; progress toward the goal without reaching it = -1 ; expected level after treatment = 0 ; "most likely" level after treatment = +1 ; successful goal better than expected = +2]
Motor imagery capability | Day-30 ; Day 90 ; Day 180
  Motor imagery capability will be measured by the Tongue Mouth Imagery Questionnaire by the same blind and experienced physical therapist. It consists in scoring the vividness of motor imagery movement using a 5-point Likert scale separating the visual and kinesthetic modalities (1: no image/sensation, 5: image as clear / sensation as intense as during overt movement).

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Cabinet Bataille, Lyon
  - Cabinet de kinésithérapie Saint Alexandre, Lyon
  - Hôpital Henry Gabrielle, Saint-Genis-Laval

IPD SHARING:
Plan to Share IPD: No